CLINICAL TRIAL: NCT01219530
Title: Follow Up of Gestational Carriers and Intended Parents
Status: Withdrawn | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2010-01
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Attitudes; Reactions; Psychopathology
Keywords: gestational carrier; intended parent
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gestational Carriers
- Intended Parents

SUMMARY:
To explore the attitudes and reactions of gestational carriers and intended parents though their medical, pregnancy and postpartum experiences.

DETAILED DESCRIPTION:
This study will first evaluate whether there is any existing psychopathology in gestational carriers prior to their pregnancies. Second, the study will explore the gestational carriers' and intended parents' experiences including attachment with quantitative measurements. These measurements will be collected prospectively.

ELIGIBILITY:
None, other than being either a gestational carrier or intended parent.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients participating in the gestational carrier program, either as a gestation carrier or an intended parent.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Braverman, PhD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Morristown, New Jersey, United States